CLINICAL TRIAL: NCT04875559
Title: Multimodal Pain Treatment for Breast Cancer Surgery - a Prospective Cohort Study
Status: Completed | Type: Observational
Sponsor: Zealand University Hospital (Other)
Responsible Party: Sponsor
Other Study IDs: REG-028-2021
Record Dates: First submitted 2021-04-19; First posted 2021-05-06 (Actual); Last update posted 2023-07-14 (Actual); Status verified 2023-07

CONDITIONS: Breast Cancer Female; Postoperative Pain; Postoperative Nausea and Vomiting
Keywords: Multimodal pain management; Opioid-sparing pain management; Quality of recovery
MeSH Terms: conditions — Pain, Postoperative; Postoperative Nausea and Vomiting

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Patient Registry: Yes
Target Follow-Up Duration: 12 Months
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- Breast cancer surgery patients.: Patients scheduled for day-case unilateral breast conserving surgery or mastectomy with or without axillary lymph node dissection or sentinel lymph node biopsy. No intervention.
  Interventions: Other: Standardised multimodal pain treatment regimen

INTERVENTIONS:
Other: Standardised multimodal pain treatment regimen — Preoperatively:
  * Paracetamol 1000 mg p.o.
  * Celecoxib 400 mg p.o.
  * Dexamethasone 12 mg p.o.
  Perioperatively:
  * Ondansetron 4 mg IV
  * Bupivacaine 2.5 mg/mL, 20 mL LIA
  * Oxycodone 0.15 mg/kg IV (Oxycodone 0.25 mg/kg for ALND)
  Postoperatively:
  * Paracetamol 1000 mg p.o. every 6h PRN
  * Ibuprofen 400 mg p.o. every 6h (day 1-5) PRN
  * Oxycodone 5 mg IV or 10 mg p.o. PRN
  * Ondansetron 4 mg IV or p.o. PRN

SUMMARY:
Breast cancer is one of the most common types of cancer among women worldwide. (1) Breast-conserving surgery or mastectomy is indicated for the majority of patients with this type of cancer. (2) Postoperative pain is frequent in this population, with almost 50 % experiencing acute pain and 25-60 % subsequently live with chronic pain. (3-5) Today no golden standard for postoperative pain management regarding breast cancer surgeries exists, and there is definitely room for improvement. Especially considering the large population of women with breast cancer and consequences of acute and chronic pain, such as prolonged recovery and affected quality of life. (6,7) With the present study, we aim to optimise postoperative pain treatment and investigate the effect of a standardised multimodal postoperative analgesic regimen based on previous recommendations. (4,8,9)

DETAILED DESCRIPTION:
All patients scheduled for breast conserving surgery or mastectomy with or without ALND or SLNB at Zealand University Hospital, Roskilde, will be invited to participate in the study. When the patients arrive for preoperative preparation on the day of surgery, one of the investigators will be responsible for a thorough oral information regarding the purpose of the study and all relevant participation requirements. The conversation will take place in a closed room, and the informed consent form will be obtained if the patient decides to participate.

Furthermore, patients will be informed that participation is voluntary and that a wish for withdrawal will be granted immediately.

The informed consent will grant the investigators direct access to data in the patients' electronic files to ensure the information necessary for the study. The patients also consent to complete the questionnaires in the seven-day follow-up period, and that the investigators can reach them by phone.

Completion of the study It is considered a completion of the study when a patient has signed the informed consent, has followed the treatment regimen, and answered the questionnaires in the seven-day follow-up period.

If a patient does not complete the study, an account should be given as to whether and how this subject's data is handled in the study - this also replies to drop-outs.

Reasons for withdrawal

- If a patient wishes to withdraw from the study In accordance with the Declaration of Helsinki, patients have the right to withdraw from the study at any time for any reason. The investigators also have the right to withdraw a patient from the study at any time. The reason for withdrawal must be recorded.

ELIGIBILITY:
Inclusion Criteria:

* Patients scheduled for day-case unilateral breast conserving surgery or mastectomy +/- ALND or SLNB.
* Age ≥ 18 years of age.
* Patients who received written and oral information, and have signed the informed consent form on participation in the study.
* Patients living in the Region of Zealand.

Exclusion Criteria:

* Not able to speak, read, or understand Danish.
* Inability to cooperate and to consent.

Min Age: 18 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: All patients scheduled for breast conserving surgery or mastectomy with or without ALND or SLNB at Zealand University Hospital, Roskilde, will be invited to participate in the study.
Sampling Method: Probability Sample
Enrollment: 236 (Actual)
Dates: Start 2021-04-19 (Actual); Primary Completion 2022-08-04 (Actual); Study Completion 2022-08-18 (Actual)

PRIMARY OUTCOMES:
Postoperative pain | Postoperative day 1 to 7.
  Postoperative pain scored on the 11-point numeric rating scale, NRS, (score 0 = no pain, 10 = worst pain imaginable). Average pain, worst pain and pain during arm abduction to an angle of 90 degrees out from the body.

SECONDARY OUTCOMES:
Pain at the day-case post anaesthesia care unit (dcPACU) | From arrival to the dcPACU until discharged from the dcPACU, up to 5 hours
  Pain at dcPACU arrival and worst pain during dcPACU stay, scored on the 11-point numeric rating scale, NRS, (score 0 = no pain, 10 = worst pain imaginable).
Postanaesthesia recovery time | From arrival to the dcPACU until discharged from the dcPACU, up to 5 hours
  Length of stay at day-case post anaesthesia care unit (dcPACU).
Postoperative nausea and vomiting | Postoperative day 1 to 7.
  Nausea on average and at worst, measured on a four-point Likert scale (0 = none, 1 = slight, 2 = moderate, 3 = severe). Vomiting (yes/no)
Daily use of analgesics | Postoperative day 1 to 7.
  Type of drug and dosage
Location of pain | Day of surgery (preoperative) and postoperative day 1 to 7.
  Patient's perceived location of pain preoperatively and postoperatively (questionnaire options: breast, side of chest, axilla, arm)
Quality of sleep | Postoperative day 1 to 7.
  Patient's perceived quality of sleep (questionnaire options: good, difficulty of falling asleep, frequent awakenings, no sleep).
Well-being | Postoperative day 1 to 7.
  Patient's perceived feelings of sadness (yes/no), restlessness (yes/no), or fatigue (yes/no).
Quality of recovery, QoR-15D | Postoperative day 1 and 7.
  The QoR-15D is a validated questionnaire (danish version) resulting in a score of 1-150.

CONTACTS AND LOCATIONS:
Overall Officials: Anne Sofie N Therkelsen, MD, Principal Investigator — Department of Anaesthesiology, Zealand University Hospital, Roskilde, Denmark
Locations (1):
- Zealand University Hospital, Department of Anaesthesiology, Roskilde, Denmark

REFERENCES:
- [Background] Sung H, Ferlay J, Siegel RL, Laversanne M, Soerjomataram I, Jemal A, Bray F. Global Cancer Statistics 2020: GLOBOCAN Estimates of Incidence and Mortality Worldwide for 36 Cancers in 185 Countries. CA Cancer J Clin. 2021 May;71(3):209-249. doi: 10.3322/caac.21660. Epub 2021 Feb 4. PMID 33538338
- [Background] Moo TA, Sanford R, Dang C, Morrow M. Overview of Breast Cancer Therapy. PET Clin. 2018 Jul;13(3):339-354. doi: 10.1016/j.cpet.2018.02.006. PMID 30100074
- [Background] Habib AS, Kertai MD, Cooter M, Greenup RA, Hwang S. Risk factors for severe acute pain and persistent pain after surgery for breast cancer: a prospective observational study. Reg Anesth Pain Med. 2019 Feb;44(2):192-199. doi: 10.1136/rapm-2018-000040. Epub 2019 Jan 5. PMID 30700614
- [Background] Lepot A, Elia N, Tramer MR, Rehberg B. Preventing pain after breast surgery: A systematic review with meta-analyses and trial-sequential analyses. Eur J Pain. 2021 Jan;25(1):5-22. doi: 10.1002/ejp.1648. Epub 2020 Oct 4. PMID 32816362
- [Background] Gartner R, Kroman N, Callesen T, Kehlet H. Multimodal prevention of pain, nausea and vomiting after breast cancer surgery. Minerva Anestesiol. 2010 Oct;76(10):805-13. PMID 20935616
- [Background] Gong Y, Tan Q, Qin Q, Wei C. Prevalence of postmastectomy pain syndrome and associated risk factors: A large single-institution cohort study. Medicine (Baltimore). 2020 May;99(20):e19834. doi: 10.1097/MD.0000000000019834. PMID 32443289
- [Background] Sagen A, Karesen R, Sandvik L, Risberg MA. Changes in arm morbidities and health-related quality of life after breast cancer surgery - a five-year follow-up study. Acta Oncol. 2009;48(8):1111-8. doi: 10.3109/02841860903061691. PMID 19863218
- [Background] Jacobs A, Lemoine A, Joshi GP, Van de Velde M, Bonnet F; PROSPECT Working Group collaborators#. PROSPECT guideline for oncological breast surgery: a systematic review and procedure-specific postoperative pain management recommendations. Anaesthesia. 2020 May;75(5):664-673. doi: 10.1111/anae.14964. Epub 2020 Jan 26. PMID 31984479
- [Background] Steinthorsdottir KJ, Awada HN, Abildstrom H, Kroman N, Kehlet H, Aasvang EK. Dexamethasone Dose and Early Postoperative Recovery after Mastectomy: A Double-blind, Randomized Trial. Anesthesiology. 2020 Apr;132(4):678-691. doi: 10.1097/ALN.0000000000003112. PMID 31977520
- [Derived] Petersen M, Joost M, Therkelsen AS, Geisler A. Women's Experiences of Sequelae After Mastectomy: A 3, 6, and 12 Months' Follow-up Study. Cancer Nurs. 2025 Sep-Oct 01;48(5):401-408. doi: 10.1097/NCC.0000000000001341. Epub 2024 Mar 7. PMID 40838964